CLINICAL TRIAL: NCT06748846
Title: Efficacy of Segmental Muscle Vibration on Pain Modulation in Patients With Primary Cervical Dystonia: a Randomized Controlled Study
Brief Title: Segmental Muscle Vibration on Pain in Patients With Primary Cervical Dystonia
Acronym: VIBRA-DYSTONIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VIBRA-DYSTONIA
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Primary Cervical Dystonia
Keywords: Primary Cervical Dystonia; rehabilitation; Focal vibration
MeSH Terms: conditions — Cervical Dystonia, Primary | interventions — Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focal Muscle Vibration (Experimental): Patients receive 10 sessions of integrated rehabilitation, including 45 minutes of physiotherapy, 15 minutes of therapeutic Focal Muscle Vibration, and 30 minutes of occupational therapy
  Interventions: Device: Physiotherapy + Occupational therapy + Focal Muscle Vibration
- Sham Focal Muscle Vibration (Sham Comparator): Patients receive an identical protocol, but the Focal Muscle Vibration is sham (the vibration device produces sound but no actual vibration).
  Interventions: Device: Physiotherapy + Occupational therapy + Sham Focal Muscle Vibration

INTERVENTIONS:
Device: Physiotherapy + Occupational therapy + Focal Muscle Vibration — - Physiotherapy (60 minutes): Includes active strengthening of antagonist muscles, mobilization, stretching of cervical-thoracic kinetic chains, proprioceptive control, postural exercises, and body schema modulation. -Occupational Therapy (30 minutes): Focuses on improving proprioceptive, praxis, and spatial control of movements. -SMV (15 minutes): Administered during the last part of each physiotherapy session. Experimental Group: SMV is applied to the trapezius (middle/descending fibers) and quadratus lumborum bilaterally at 80 Hz with an amplitude of 0.5 mm.
  Arms: Focal Muscle Vibration
Device: Physiotherapy + Occupational therapy + Sham Focal Muscle Vibration — Physiotherapy (60 minutes): Includes active strengthening of antagonist muscles, mobilization, stretching of cervical-thoracic kinetic chains, proprioceptive control, postural exercises, and body schema modulation. Occupational Therapy (30 minutes): Focuses on improving proprioceptive, praxis, and spatial control of movements. SMV (15 minutes): Administered during the last part of each physiotherapy session. Control Group: Sham SMV using disconnected terminals produces sound but no vibration, ensuring blinding.
  Arms: Sham Focal Muscle Vibration

SUMMARY:
This pilot study aims to evaluate the effectiveness of Vibration Muscle Stimulation (VMS) in reducing pain and improving quality of life in patients with primary cervical dystonia (CD), a focal dystonia characterized by involuntary and often painful muscle contractions in the neck. The study will involve patients who have been treated with botulinum toxin and are candidates for an integrated rehabilitation program, which includes physiotherapy and occupational therapy. Participants will be randomized into two groups: an experimental group receiving therapeutic VMS (80 Hz frequency, 0.5 mm vibration amplitude) and a control group receiving sham VMS. Both groups will undergo a 10-session rehabilitation program combining 45 minutes of physiotherapy and 15 minutes of VMS (or sham), followed by 30 minutes of occupational therapy. The primary outcome measure will be pain and disability as assessed by the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) and the McGill Pain Questionnaire. Secondary outcomes will include improvements in quality of life and clinical severity of dystonia. The results are expected to provide insights into the potential role of VMS in enhancing rehabilitation outcomes for patients with cervical dystonia.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of Vibration Muscle Stimulation (VMS) in reducing pain and improving quality of life in patients with primary cervical dystonia (CD), a focal dystonia characterized by involuntary and often painful muscle contractions in the neck. The study will involve patients who have been treated with botulinum toxin and are candidates for an integrated rehabilitation program, which includes physiotherapy and occupational therapy. Participants will be randomized into two groups: an experimental group receiving therapeutic VMS (80 Hz frequency, 0.5 mm vibration amplitude) and a control group receiving sham VMS. Both groups will undergo a 10-session rehabilitation program combining 45 minutes of physiotherapy and 15 minutes of VMS (or sham), followed by 30 minutes of occupational therapy. The primary outcome measure will be pain and disability as assessed by the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) and the McGill Pain Questionnaire. Secondary outcomes will include improvements in quality of life and clinical severity of dystonia. The results are expected to provide insights into the potential role of VMS in enhancing rehabilitation outcomes for patients with cervical dystonia.

Detailed Description This study aims to evaluate the efficacy of Segmental Muscle Vibration (SMV) on pain reduction and quality of life improvement in patients with primary cervical dystonia (CD). The study is conducted on patients undergoing botulinum toxin treatment and eligible for a standardized integrated rehabilitation protocol, including physiotherapy and occupational therapy. Cervical dystonia is a neurological disorder characterized by involuntary contractions of neck muscles, leading to abnormal movements, postures, and significant pain. Current treatment often involves botulinum toxin injections, but additional therapeutic strategies are required to address persistent symptoms such as pain and impaired quality of life. SMV, a non-invasive intervention, applies mechanical vibration to specific muscles to modulate pain perception, improve proprioception, and enhance motor function. This study seeks to determine the translational potential of SMV as a component of integrated rehabilitation in CD patients.

The study is a single-center, randomized controlled trial with parallel arms. Patients in the experimental group will receive 10 sessions of integrated rehabilitation, including 45 minutes of physiotherapy, 15 minutes of therapeutic SMV, and 30 minutes of occupational therapy. Patients in the control group will follow an identical protocol, but the SMV will be sham (the vibration device produces sound but no actual vibration). Participants are recruited from the Spasticity Outpatient Clinic at Fondazione Don Gnocchi, Rovato (BS), Italy, where they are treated for painful cervical dystonia with botulinum toxin. After receiving the toxin, patients meeting inclusion criteria are briefed on the study's purpose and procedures. Upon signing informed consent, participants undergo an initial evaluation (T0) by a physiatrist, who assigns them randomly to either the experimental or control group using a pre-sealed envelope system.

The rehabilitation program consists of 10 outpatient sessions. Each session includes physiotherapy for 60 minutes, which involves active strengthening of antagonist muscles, mobilization, stretching of cervical-thoracic kinetic chains, proprioceptive control, postural exercises, and body schema modulation. Occupational therapy follows for 30 minutes, focusing on improving proprioceptive, praxis, and spatial control of movements. SMV is administered during the last part of each physiotherapy session. In the experimental group, SMV is applied to the trapezius (middle/descending fibers) and quadratus lumborum bilaterally at 80 Hz with an amplitude of 0.5 mm. In the control group, sham SMV is applied using disconnected terminals that produce sound but no vibration, ensuring blinding.

Participants will be evaluated at baseline (T0), after five sessions (T1), and after completing the program (T2) using standardized scales. The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) will assess clinical severity, disability, and pain. The McGill Pain Questionnaire will evaluate pain perception and subjective experience. The Tsui Score will measure the clinical severity of dystonia, including amplitude and duration of dystonic movements, tremor, and shoulder elevation. Randomization is performed using sequentially numbered, sealed envelopes containing group allocation. Both patients and therapists are blinded to the group assignment, and sham SMV mimics the sound of active SMV without delivering vibration.

Participants will undergo 10 sessions over 5 weeks, with evaluations occurring at three time points: T0 (pre-treatment, baseline), T1 (mid-treatment, after 5 sessions), and T2 (post-treatment, after 10 sessions). The same evaluator will administer the scales across all time points to ensure consistency. This study aims to establish SMV as a non-invasive, adjunctive treatment option for cervical dystonia, targeting pain relief and improved functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary cervical dystonia.
* Pain intensity >3 on the Numerical Rating Scale (NRS).
* Recent botulinum toxin therapy (within 30 days).
* Age ≥18 years.
* MMSE >24 (no significant cognitive impairment).

Exclusion Criteria:

* Non-ambulatory status.
* Generalized dystonia or non-cervical forms.
* Inflammatory, neurodegenerative, or rheumatological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) | From enrollment to the end of treatment at 5 weeks
  Assesses clinical severity, disability, and pain.
McGill Pain Questionnaire | From enrollment to the end of treatment at 5 weeks
  Evaluates pain perception and subjective experience.

SECONDARY OUTCOMES:
Tsui Score Measures | From enrollment to the end of treatment at 5 weeks
  The clinical severity of dystonia, including amplitude and duration of dystonic movements, tremor, and shoulder elevation.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Fondazione Don Gnocchi "E. Spalenza", Rovato, Brescia, Italy

REFERENCES:
- [Result] Tijssen MA, Marsden JF, Brown P. Frequency analysis of EMG activity in patients with idiopathic torticollis. Brain. 2000 Apr;123 ( Pt 4):677-86. doi: 10.1093/brain/123.4.677. PMID 10733999
- [Derived] Buraschi R, Pedersini P, Redegalli G, Pullara R, Pollet J, Rossi M, Gobbo M, Gueli S, Falso M. Efficacy of Segmental Muscle Vibration on Pain Modulation in Patients with Primary Cervical Dystonia Treated with Botulinum Type-A Toxin: A Protocol for a Randomized Controlled Trial. NeuroSci. 2025 Apr 2;6(2):30. doi: 10.3390/neurosci6020030. PMID 40265360